CLINICAL TRIAL: NCT07375186
Title: Comparison of Oral Carbohydrate Solution Versus Clear Liquid Diet in Acute Pancreatitis:A Randomized Controlled Trial
Brief Title: Early Oral Carbohydrate Solution vs Clear Liquid Diet in Acute Pancreatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Hospital (Other)
Responsible Party: Principal Investigator, Aiqa Gulshan, Resident Surgeon, Jinnah Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERB198/07/01-0-1-2026/AIMC/JHL
Record Dates: First submitted 2026-01-03; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Acute Pancreatitis
Keywords: Oral Carbohydrates in Acute Pancreatitis; Early feeding choice in Acute Pancreatitis; Clear liquid diet in Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORAL CARBOHYDRATE SOLUTION GROUOP (Experimental): Participant will be randomized in this group. Participant will receive an oral carbohydrate solution initiated after clinical stabilization.It will be be administrated orally with volume and frequency standardized for all participants and advancement according to study protocol.
  Interventions: Dietary Supplement: Oral Carbohydrate Solution
- CLEAR LIQUID DIET GROUP (Active Comparator): Participant will receive a standard clear liquid diet initiated after clinical stabilization as per routine institutional practice in measured frequncy and volume and advancement according to study protocol.
  Interventions: Dietary Supplement: Clear Liquid diet

INTERVENTIONS:
Dietary Supplement: Oral Carbohydrate Solution — Participant will be allocated in oral carbohydrate solution group.Participant will receive an oral carbohydrate solution initiated after clinical stabilization.It will be be administrated orally with volume and frequency standardized for all participants and advancement according to study protocol.
  Arms: ORAL CARBOHYDRATE SOLUTION GROUOP
Dietary Supplement: Clear Liquid diet — Participant will receive a standard clear liquid diet initiated after clinical stabilization as per routine institutional practice in measured frequncy and volume and advancement according to study protocol.
  Arms: CLEAR LIQUID DIET GROUP

SUMMARY:
Background:

Acute pancreatitis (AP) is an inflammatory condition associated with increased metabolic demands and negative nitrogen balance, making early nutritional support a critical component of management. Concentional practice favored prolonged fasting and delayed oral intake; however, recent evidence supports early oral feeding. Oral carbohydrate solutions (OCS) may provide early caloric support with minimal pancreatic stimulation, but data comparing OCS with clear liquid (CL) diets which is current practice remain limited, particularly in South Asian populations.The Convential diet (CD )group started at liquid diet then progressed towards soft and then solid diet experienced recurring pain at a considerably higher rate than the oral high carbohydrate solution (OCS )group providing essential calories,(13.2% vs. 3.8%, p < 0.001).OCS showed decrease rate of post prandial recurrent abdominal pain.

Objective:

To compare oral carbohydrate solution versus clear liquid diet as the initial oral feeding strategy in patients with acute pancreatitis, focusing on feeding intolerance and length of hospital stay.

Methods:

This prospective randomized controlled trial will be conducted at a tertiary-care hospital in Lahore, Pakistan. Adult patients (18-70 years) with mild to moderately severe acute pancreatitis will be randomized to receive either an oral carbohydrate solution (10% dextrose in water) or a clear liquid diet as the initial oral feed. The primary outcomes will be feeding intolerance within 24 hours and length of hospital stay. Secondary outcomes include time to successful oral feeding, time to soft diet, changes in pain scores, inflammatory markers (CRP, WBC), glycemic response, need for nutritional escalation, complications, and patient satisfaction. Data will be analyzed using SPSS version 26, with a p-value ≤ 0.05 considered statistically significant.

Conclusion:

If proven safe and effective, oral carbohydrate solution may serve as a simple, cost-effective and well-tolerated alternative to clear liquid diets for early oral feeding in acute pancreatitis, particularly in resource limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 years and 70 years
* Diagnosis of mild or moderately severe acute pancreatitis
* Hemodynamically stable
* Able to tolerate oral intake
* Provided written informed consent

Exclusion Criteria:

* Severe acute pancreatitis
* Chronic pancreatitis
* Pregnancy
* Uncontrolled diabetes mellitus
* Known malabsorption syndrome,
* Patients requiring immediate enteral tube feeding or parenteral nutrition,
* Known allergy or intolerance to carbohydrate solutions,
* Persistent retching or vomiting

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
rate of feeding intolerance | Upto 24 hours after initiating first oral feed
  Patient will be observed for 24 hours after initial feed for symptoms of feeding intolerance like pain,nausea,vomiting or abdominal distension.
Length of hospital Stay | From hospital admission to discharge in days
  Length of hospital stay will be recorded from day of admission till discharge in days.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan